CLINICAL TRIAL: NCT05928455
Title: A Clinical Trial to Assess the Immunogenicity and Safety Following a Heterologous Booster Dose of Recombinant SARS-CoV-2 Vaccine (CHO Cell) LYB001 in Adults 18-59 Years of Age Completed Two- or Three-dose Inactivated COVID-19 Vaccine
Brief Title: The Immunogenicity and Safety Following a Heterologous Booster Dose of Recombinant SARS-CoV-2 Vaccine LYB001
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangzhou Patronus Biotech Co., Ltd. (Industry)
Collaborators: Yantai Patronus Biotech Co., Ltd. (Industry); Afﬁliated Hospital of North Sichuan Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MLD-C-22001
Record Dates: First submitted 2023-06-21; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: COVID-19; Vaccine Reaction
Keywords: Safety; immunogenicity; heterologous booster; inactivated COVID-19 vaccine; recombinant SARS-CoV-2 vaccine
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Randomized, open label, positive control (Stage Ⅰ); Single-arm, open-label (Stage Ⅱ)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LYB001 (Experimental): Participants receiving a boost with 30ug or 60ug LYB001 after a two-or three-dose primary series of inactivated COVID-19 vaccine.
  Interventions: Biological: LYB001
- CoronaVac (Active Comparator): Participants receiving a boost with vaccine CoronaVac after a two-or three-dose primary series of inactivated COVID-19 vaccine.
  Interventions: Biological: CoronaVac

INTERVENTIONS:
Biological: LYB001 — Experimental: The LYB001 vaccine was administered through intramuscular injection at doses of 30ug or 60ug in a 0.5mL volume.
  Arms: LYB001
Biological: CoronaVac — Active Comparator: The CoronaVac vaccine was administered through intramuscular injection in a 0.5mL volume.
  Arms: CoronaVac

SUMMARY:
The goal of this clinical trial is to assess the immunogenicity and safety following a heterologous booster dose of recombinant SARS-CoV-2 vaccine (CHO cell) LYB001 in adults 18-59 years of age completed two- or three-dose inactivated COVID-19 vaccine. The main questions it aims to answer are:

* whether LYB001 group is better on immunogenicity than the control group of inactivated vaccine?
* whether LYB001 group has better performance on safety than the control group of inactivated vaccine, such as the lower adverse reaction rate?

DETAILED DESCRIPTION:
Primary Objectives

1. To assess the immunogenicity profile following a heterologous booster dose of LYB001 as compared to a homologous booster dose of inactivated vaccine in adults 18-59 years of age completed two- or three-dose primary series of inactivated vaccine.
2. To assess the safety profile following a heterologous booster dose of LYB001 as compared to a homologous booster dose of inactivated vaccine in adults 18-59 years of age completed two- or three-dose primary series of inactivated vaccine.

Secondary Objectives 1) To assess the immune durability following a heterologous booster dose of LYB001 as compared to a homologous booster dose of inactivated vaccine in adults 18-59 years of age completed two- or three-dose primary series of inactivated vaccine.

Exploratory objectives

1) To assess the cellular immune response following a heterologous booster dose of LYB001 as compared to a homologous booster dose of inactivated vaccine in adults 18-59 years of age completed two- or three-dose primary series of inactivated vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged 18-59 years, including both males and females;
2. Subjects who agree to participate in this clinical trial voluntarily and sign the informed consent form, are capable of providing valid identification, understanding and complying with the requirements of the clinical protocol.
3. Subjects who have completed two- or three-dose inactivated COVID-19 vaccine at 6-12 months earlier.
4. For female participants of childbearing potential, effective contraception measures should be used within 2 weeks prior to participation in this study and the results of pregnancy test is required to be negative. Participants should voluntarily agree to use effective contraceptive measures from the time of signing the informed consent form to the end of the study (effective contraceptive measures including oral contraceptives (excluding emergency contraceptives), injectable or implantable contraceptives, sustained-release topical contraceptives, hormonal patches, intrauterine device, sterilization, abstinence, condoms (for males), diaphragms, cervical caps, etc.).

Exclusion Criteria:

1. Receipt of any COVID-19 prophylactic medication (e.g., receipt history of any approved or under developing COVID-19 vaccines other than inactivated vaccine), or previous vaccination history other than other than two or three doses of inactivated vaccination;
2. Abnormal vital signs with clinical significance prior to enrolment, with systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, or axillary body temperature ≥ 37.3°C prior to enrolment; abnormal results of laboratory screening tests which was clinically significant judged by clinicians prior to enrolment.
3. Known allergy, or history of anaphylaxis or other serious adverse reactions to vaccines or their excipients;
4. History of severe acute respiratory syndrome (SARS) or Middle East respiratory syndrome (MERS);
5. History of COVID-19, or history of close contact with confirmed/suspected COVID-19 patients, or positive results for SARS-CoV-2 nucleic acid tests at screening;
6. Administration of antipyretics, painkillers or anti-allergy drugs within 24 hours prior to enrolment;
7. Receipt of any live attenuated vaccine within 28 days prior to vaccination and other vaccines, such as subunit and inactivated vaccine within 14 days prior to vaccination;
8. Receipt of blood or blood-related products, including immunoglobulins, within 3 months prior to vaccination; or any planned use during the study period.
9. Subjects with the following diseases:

   1. Any acute diseases or acute attacks of chronic diseases within 7 days prior to enrolment；
   2. Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.；
   3. Congenital or acquired immunodeficiency or autoimmune disease, or long-term receipt (>14 consecutive days) of glucocorticoid (reference value for dose: ≥20 mg/day prednisone or equivalent) or other immunosuppressive agents within the past 6 months, with exception of inhaled or topical steroids, or short-term use (≤14 consecutive days) of oral corticosteroids；
   4. Currently suffering from or diagnosed with infectious diseases, positive screening results for hepatitis B surface antigen, hepatitis C antibody, treponema pallidum antibody, human immunodeficiency virus antibody；
   5. History or family history of neurological disorders (convulsions, epilepsy, encephalopathy, etc.) or psychiatric disorders；
   6. Asplenia, or functional asplenia；
   7. Presence of severe, uncontrollable or hospitalized cardiovascular diseases, diabetes, blood and lymphatic diseases, immune diseases, liver and kidney diseases, respiratory diseases, metabolic and skeletal diseases, or malignant tumors;
   8. Contraindications to IM injections and blood draws, such as coagulation disorders, thrombotic or bleeding disorders, or conditions that needs continuous anticoagulant usage.
10. Drug or alcohol abuse (alcohol intake ≥ 14 units per week) which in the investigator's opinion would compromise the participant's safety or compliance with the study procedures;
11. Pregnant or lactating females;
12. Having participated or participating in COVID-19 related clinical trials, and those participating or planning to participate in other clinical trials during the study period;
13. Presence of any underlying disease or condition which, in the opinion of the investigator, may place the subject at unacceptable risk, is unable to meet the requirements of the protocol, or interfere with the assessment of vaccine response.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-05-14 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The Seroconversion (SCRs) of neutralizing antibodies (Nabs) and S protein-binding antibodies at 14 days after the booster immunization | 14 days after booster vaccination
  The Seroconversion (SCRs) with Clopper-Pearson 95% CIs of neutralizing antibodies (Nabs) against prototype SARS-CoV-2 and circulating VOCs using Vesicular stomatitis virus (VSV)-based pseudovirus neutralizing assays, S protein-binding antibodies using ELISA assays, at 14 days after the booster immunization will be calculated for each group, respectively.
The Seroconversion (SCRs) of neutralizing antibodies (Nabs) and S protein-binding antibodies at 28 days after the booster immunization | 28 days after booster vaccination
  The Seroconversion (SCRs) with Clopper-Pearson 95% CIs of neutralizing antibodies (Nabs) against prototype SARS-CoV-2 and circulating VOCs using Vesicular stomatitis virus (VSV)-based pseudovirus neutralizing assays, S protein-binding antibodies using ELISA assays, at 28 days after the booster immunization will be calculated for each group, respectively.
The Geometric Neutralizing titers (GMT) of neutralizing antibodies (Nabs) and S protein-binding antibodies at 14 days after booster vaccination | 14 days after booster vaccination
  The Geometric Neutralizing titers (GMT) with Clopper-Pearson 95% CIs of neutralizing antibodies (Nabs) against prototype SARS-CoV-2 and circulating VOCs using Vesicular stomatitis virus (VSV)-based pseudovirus neutralizing assays, S protein-binding antibodies using ELISA assays, at 14 days after the booster immunization will be calculated for each group, respectively.
The Geometric Neutralizing titers (GMT) of neutralizing antibodies (Nabs) and S protein-binding antibodies at 28 days after booster vaccination | 28 days after booster vaccination
  The Geometric Neutralizing titers (GMT) with Clopper-Pearson 95% CIs of neutralizing antibodies (Nabs) against prototype SARS-CoV-2 and circulating VOCs using Vesicular stomatitis virus (VSV)-based pseudovirus neutralizing assays, S protein-binding antibodies using ELISA assays, at 28 days after the booster immunization will be calculated for each group, respectively.
The Geometric mean fold rise (GMFR) of neutralizing antibodies (Nabs) and S protein-binding antibodies at 14 days after the booster immunization compared with the baseline | 14 days after booster vaccination
  The Geometric mean fold rise (GMFR) with Clopper-Pearson 95% CIs of neutralizing antibodies (Nabs) against prototype SARS-CoV-2 and circulating VOCs using Vesicular stomatitis virus (VSV)-based pseudovirus neutralizing assays, S protein-binding antibodies using ELISA assays, at 14 days after the booster immunization will be calculated for each group, compared with the baseline, respectively.
The Geometric mean fold rise (GMFR) of neutralizing antibodies (Nabs) and S protein-binding antibodies at 28 days after the booster immunization compared with the baseline | 28 days after booster vaccination
  The Geometric mean fold rise (GMFR) with Clopper-Pearson 95% CIs of neutralizing antibodies (Nabs) against prototype SARS-CoV-2 and circulating VOCs using Vesicular stomatitis virus (VSV)-based pseudovirus neutralizing assays, S protein-binding antibodies using ELISA assays, at 28 days after the booster immunization will be calculated for each group, compared with the baseline, respectively.
The frequencies and percentages of adverse events within 30 minutes after booster vaccination | within 30 minutes after booster vaccination
  Statistical description of solicited and unsolicited adverse events (AEs) will be listed. Frequencies and percentages of AEs, including overall AEs, AEs related to vaccination, AEs classified as grade 3 or worse, AEs classified as grade 3 or worse that related to vaccination, AEs leading to participant's withdrawal, AEs leading to participant's withdrawal that related to vaccination will be presented. Fisher's exact test will be used to compare the differences between the groups.
  Solicited and unsolicited AEs within 30 mins after vaccination will be collected.
The frequencies and percentages of adverse events within 7 days after booster vaccination | within 7 days after booster vaccination
  Statistical description of solicited and unsolicited adverse events (AEs) will be listed. Frequencies and percentages of AEs, including overall AEs, AEs related to vaccination, AEs classified as grade 3 or worse, AEs classified as grade 3 or worse that related to vaccination, AEs leading to participant's withdrawal, AEs leading to participant's withdrawal that related to vaccination will be presented. Fisher's exact test will be used to compare the differences between the groups.
  Solicited and unsolicited AEs within 7 days after vaccination will be collected.
The frequencies and percentages of unsolicitedadverse events within 8-28 days after booster vaccination | within 8-28 days after booster vaccination
  Statistical description of solicited and unsolicited adverse events (AEs) will be listed. Frequencies and percentages of AEs, including overall AEs, AEs related to vaccination, AEs classified as grade 3 or worse, AEs classified as grade 3 or worse that related to vaccination, AEs leading to participant's withdrawal, AEs leading to participant's withdrawal that related to vaccination will be presented. Fisher's exact test will be used to compare the differences between the groups.
  Unsolicited AEs within 8-28 days after vaccination will be collected.

SECONDARY OUTCOMES:
The Seroconversion (SCRs) of neutralizing antibodies (Nabs) and S protein-binding at 3 months after booster vaccination | 3 months after booster vaccination
  The Seroconversion (SCRs) with Clopper-Pearson 95% CIs of NAbs against prototype SARS-CoV-2 and circulating VOCs, S protein-binding antibodies, at 3 months after booster vaccination will be calculated for each group, respectively.
The Seroconversion (SCRs) of neutralizing antibodies (Nabs) and S protein-binding at 6 months after booster vaccination | 6 months after booster vaccination
  The Seroconversion (SCRs) with Clopper-Pearson 95% CIs of NAbs against prototype SARS-CoV-2 and circulating VOCs, S protein-binding antibodies, at 6 months after booster vaccination will be calculated for each group, respectively.
The Seroconversion (SCRs) of neutralizing antibodies (Nabs) and S protein-binding at 12 months after booster vaccination | 12 months after booster vaccination
  The Seroconversion (SCRs) with Clopper-Pearson 95% CIs of NAbs against prototype SARS-CoV-2 and circulating VOCs, S protein-binding antibodies, at 12 months after booster vaccination will be calculated for each group, respectively.
The Geometric Neutralizing titers (GMT) of neutralizing antibodies (Nabs) and S protein-binding antibodies at 3 months after booster vaccination | 3 months after booster vaccination
  The Geometric Neutralizing titers (GMT) with Clopper-Pearson 95% CIs of NAbs against prototype SARS-CoV-2 and circulating VOCs, S protein-binding antibodies, at 3 months after booster vaccination will be calculated for each group, respectively.
The Geometric Neutralizing titers (GMT) of neutralizing antibodies (Nabs) and S protein-binding antibodies at 6 months after booster vaccination | 6 months after booster vaccination
  The Geometric Neutralizing titers (GMT) with Clopper-Pearson 95% CIs of NAbs against prototype SARS-CoV-2 and circulating VOCs, S protein-binding antibodies, at 6 months after booster vaccination will be calculated for each group, respectively.
The Geometric Neutralizing titers (GMT) of neutralizing antibodies (Nabs) and S protein-binding antibodies at 12 months after booster vaccination | 12 months after booster vaccination
  The Geometric Neutralizing titers (GMT) with Clopper-Pearson 95% CIs of NAbs against prototype SARS-CoV-2 and circulating VOCs, S protein-binding antibodies, at 12 months after booster vaccination will be calculated for each group, respectively.
The Geometric mean fold rise (GMFR) of neutralizing antibodies (Nabs) and S protein-binding antibodies at 3 months after booster vaccination compared with the baseline | 3 months after booster vaccination
  The Geometric mean fold rise (GMFR) with Clopper-Pearson 95% CIs of NAbs against prototype SARS-CoV-2 and circulating VOCs, S protein-binding antibodies, at 3 months after booster vaccination will be calculated for each group, compared with the baseline, respectively.
The Geometric mean fold rise (GMFR) of neutralizing antibodies (Nabs) and S protein-binding antibodies at 6 months after booster vaccination compared with the baseline | 6 months after booster vaccination
  The Geometric mean fold rise (GMFR) with Clopper-Pearson 95% CIs of NAbs against prototype SARS-CoV-2 and circulating VOCs, S protein-binding antibodies, at 6 months after booster vaccination will be calculated for each group, compared with the baseline, respectively.
The Geometric mean fold rise (GMFR) of neutralizing antibodies (Nabs) and S protein-binding antibodies at 12 months after booster vaccination compared with the baseline | 12 months after booster vaccination
  The Geometric mean fold rise (GMFR) with Clopper-Pearson 95% CIs of NAbs against prototype SARS-CoV-2 and circulating VOCs, S protein-binding antibodies, at 12 months after booster vaccination will be calculated for each group, compared with the baseline, respectively.

OTHER OUTCOMES:
The counts of spot forming cells (SFCs) per 3×105 peripheral blood mononuclear cells (PBMCs) at 14 days after booster vaccination | 14 days after booster vaccination
  The cellular immune responses (e.g., cytokine profiling) and their changes from baseline will be statistically analysed for each group at 14 days after booster vaccination, respectively, and the differences will be statistically tested by non-parametric test.
  The cellular immune response was detected using enzyme-linked immunospot (ELISpot) assay, and presented as the counts of spot forming cells (SFCs) per 3×105 peripheral blood mononuclear cells (PBMCs) secreting interferon (IFN)-γ, interleukin (IL)-2, IL-4 when stimulated by the antigen peptide pool ex vivo.
The counts of spot forming cells (SFCs) per 3×105 peripheral blood mononuclear cells (PBMCs) at 180 days after booster vaccination | 180 days after booster vaccination
  The cellular immune responses (e.g., cytokine profiling) and their changes from baseline will be statistically analysed for each group at 180 days after booster vaccination, respectively, and the differences will be statistically tested by non-parametric test.
  The cellular immune response was detected using enzyme-linked immunospot (ELISpot) assay, and presented as the counts of spot forming cells (SFCs) per 3×105 peripheral blood mononuclear cells (PBMCs) secreting interferon (IFN)-γ, interleukin (IL)-2, IL-4 when stimulated by the antigen peptide pool ex vivo.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolan Yong, Bachelor, Principal Investigator — Chengdu Xinhua Hospital Affiliated to North Sichuan Medical College, Chengdu, China
Locations (1):
- Chengdu Xinhua Hospital Affiliated to North Sichuan Medical College, Chengdu, Sichuan, China